CLINICAL TRIAL: NCT04228107
Title: Treatment Phenotypes for Adolescents With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-1861
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Asthma in Children; Adherence, Treatment
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — Drug Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cohort (Experimental): Participants will be enrolled in medication use monitoring. Their medication use patterns will be available to themselves and their guardians via a smartphone application, and to their asthma care providers via a portal. There will be no interventions to change medication use patterns. A portion of them will be asked to participate in a semistructured interview during which they will be asked questions about their perception of their asthma, health beliefs regarding medication use, and what they feel would be the most helpful to get them to take their asthma medicines.
  Additionally a small group of healthcare providers will be asked to participate in a focus group to collect qualitative data on medication use barriers and facilitators
  Interventions: Device: Medication monitoring

INTERVENTIONS:
Device: Medication monitoring — This is an observational study of medication use patterns. The propeller health device has reminders for controller medication use and gives feedback regarding medication use to the participant, their guardian and their asthma provider

SUMMARY:
This study will evaluate how adolescents take their asthma medications using an electronic medication monitor.

DETAILED DESCRIPTION:
This study will look at how adolescents use both their controller and rescue medications using an electronic medication monitoring platform, for the period of one year. Participants will be enrolled in a medication monitoring platform, and their asthma care provider will have access to medication usage information. The study team will collect data on medication use patterns in a real world setting for 12 months per participant. Additionally, healthcare providers will be enrolled in focus groups to determine barriers and facilitators to optimal medication use for their patients.

ELIGIBILITY:
For adolescent participants:

Inclusion Criteria:

* Diagnosis of asthma On an inhaled controller and rescue medication for which a propeller health device is available

Exclusion Criteria:

* Other significant chronic lung disease (from problem list)

  * Cystic fibrosis
  * Chronic respiratory failure
  * Tracheostomy status
  * Intersititial lung disease
* Significant developmental delay
* Taking more than 3 asthma related medications
* Primary language other than English, Spanish, Catalan, Dutch, French, German or Italian

Healthcare providers will be recruited as well to participate in focus groups as part of specific aim 2.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather EH De Keyser, MD MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 adolescent participants were enrolled for the primary aim. 10 healthcare providers were enrolled to participate in focus groups.
Groups:
- Adolescents With Medication Monitoring: Participants will be enrolled in medication use monitoring. Their medication use patterns will be available to themselves and their guardians via a smartphone application, and to their asthma care providers via a portal. There will be no interventions to change medication use patterns.
- Healthcare Provider Focus Groups: Healthcare providers will be enrolled in focus groups to discuss medication adherence in teens. Healthcare provider demographics were not collected as part of focus group participation.
Period: Overall Study
Arm/Group | Adolescents With Medication Monitoring | Healthcare Provider Focus Groups
Started | 70 | 10
Completed a Qualitative Semistructured Interview (Subset) | 21 | 0
Completed | 43 (Completed 11+ months of controller and rescue medication monitoring) | 10
Not Completed | 27 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Lost to Follow-up | 18 | 0
Not completed — No controller use data | 1 | 0
Not completed — No medication data collected | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only adolescent participants with greater than 11 months (47 weeks) of synced data were included in the final analysis.
  10 healthcare providers were enrolled for focus group participation, however demographic data was not collected on these providers.
Groups:
- Adolescents: Teens enrolled for electronic medication monitoring. 43 participants completed at least 11 months of medication monitoring and were included in the final analysis
Arm/Group | Adolescents
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only participants with greater than 11 months (47 weeks) of synced data were included in the final analysis. Those not included had less than 47 weeks of data synced from the sensors.
  years | 13.8 (1.34)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only participants with greater than 11 months (47 weeks) of synced data were included in the final analysis. Those not included had less than 47 weeks of data synced from the sensors.
  Participants
    Female | 14
    Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only participants with greater than 11 months (47 weeks) of synced data were included in the final analysis. Those not included had less than 47 weeks of data synced from the sensors.
  Participants
    Hispanic or Latino | 21
    Not Hispanic or Latino | 21
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only participants with greater than 11 months (47 weeks) of synced data were included in the final analysis. Those not included had less than 47 weeks of data synced from the sensors.
  Participants
    American Indian or Alaska Native | 1
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 5
    White | 25
    More than one race | 2
    Unknown or Not Reported | 9
FEV1 Z score [Median (Inter-Quartile Range); unit: Z score] — FEV1 Z score was directly obtained from the medical record (i.e. it is calculated based on population level characteristics and is reported as a clinical measure). Z scores of +/- 1.64 are considered within normal limits. Z scores less than -1.64 or greater than +1.64 are considered abnormal. Z scores of 0 represent the population mean. Population: Only participants with greater than 11 months (47 weeks) of synced data were included in the final analysis. Those not included had less than 47 weeks of data synced from the sensors.
  Z score | 0.18 [-0.78 to 0.8]

OUTCOME MEASURES:

1. Primary Outcome: Treatment Phenotypes
Description: The Investigators will calculate the number of participants that fall into the following treatment phenotypes: "Well controlled-good adherence", "Well controlled-poor adherence", "Poorly controlled-good adherence", "Poorly controlled-poor adherence".
  We had initially planned to report only these 4 groups, however there was a very clear breakdown into 9 groups-as we needed to consider a moderately controlled group and a moderately adherent group. Therefore the groups are reported as follows:
  Poor Adhrence, Poor control Poor adherence, moderate control poor adherence, good control
  Moderate adherence, poor control moderate adherence, moderate control moderate adherence, good control
  good adherence, poor control good adherence, moderate control good adherence, good control
  The investigators will use group based trajectory modeling to evaluate adherence and control phenotypes
Time Frame: 12 months
Measure: Number; unit: Participants
Groups:
- Adolescents: Adolescents enrolled in 1 year of electronic medication monitoring. During the study, participants had less than 1 year of data completed from the sensors for a number of reasons (most often that their device stopped syncing with the app and we were unable to re-establish a connection). Only participants with greater than 11 months of data collected were included in the final analysis. N=25 participants were excluded from the final analysis for not having a full 11+ months worth of data. Therefore the final analytic population was 45 participants.
Arm/Group | Adolescents
Number analyzed (Participants) | 43
Participants
  Poor adherence, good control | 7
  poor adherence, poor control | 2
  Moderate adherence, good control | 10
  moderate adherence, poor control | 5
  high adherence, good control | 16
  high adherence, poor control | 3

2. Secondary Outcome: Qualitative Information Regarding Barriers for Medication Use
Description: Qualitative data (semistructured interviews with patients regarding barriers to medication use.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Adolescent Interviews: Subset of adolescents who completed semistructured interviews
Arm/Group | Adolescent Interviews
Number analyzed (Participants) | 21
Participants
  Theme: poor routine | 8
  Theme: forget | 3

3. Secondary Outcome: Qualitative Information Regarding Facilitators for Medication Use
Description: Qualitative data (semistructured interviews with adolescents) regarding barriers to medication use.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescent Interviews
Number analyzed (Participants) | 21
Participants
  Theme: habit | 7
  Theme: parental reminders | 8
  Theme: good routine | 12

4. Secondary Outcome: Qualitative Information Regarding Facilitators for Medication Use
Description: Qualitative data (focus groups with healthcare providers) to determine facilitators to medication use.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Provider Focus Groups: Healthcare providers were interviewed in focus groups to evaluate their perceived barriers and facilitators to adequate medication adherence
Arm/Group | Provider Focus Groups
Number analyzed (Participants) | 10
Participants
  Theme: buy in from patient/family | 5
  Theme: tailored approach | 7

5. Secondary Outcome: Qualitative Information Regarding Barriers for Medication Use
Description: Qualitative data (focus groups with healthcare providers) to determine facilitators to medication use.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Provider Focus Groups
Number analyzed (Participants) | 10
Participants
  Theme: lack of parental involvement or parenting challenges | 5
  Theme: insurance/cost barriers | 5
  Theme: lack of adolescent understanding or prioritization | 7

ADVERSE EVENTS:
Time Frame: n/a-study was observational so adverse events were not recorded.
Groups:
- Adolescents: Adolescents monitored for medication use
Arm/Group | Adolescents
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
There were a few limitations to this evaluation. First, we were under our recruitment target. This was due to a number of factors, most importantly that most of the primary study recruitment efforts occurred during the early years of the COVID pandemic, which made recruitment challenging. Additionally, though we made every effort to ensure that study sensors remained on the participants medications, we had some participants whose devices stopped syncing at some point during analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT04228107/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT04228107/ICF_002.pdf